CLINICAL TRIAL: NCT00685880
Title: Randomized, Double Blind Comparison Trial of Prolotherapy (Dextrose) Compared to Corticosteroid Injection for the Treatment of Symptomatic Thumb Carpo-metacarpal Joint Arthritis
Brief Title: Prolotherapy Versus Steroids for Thumb Carpo-metacarpal Joint Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit adequate numbers of patients
Sponsor: Mayo Clinic (Other)
Responsible Party: Michael Joseph Gruba M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-006348
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-07

CONDITIONS: Thumb Carpometacarpal Joint Osteoarthritis
Keywords: thumb carpo metacarpal joint osteoarthritis; prolotherapy; intra articular steroid; hand therapy
MeSH Terms: interventions — Prolotherapy; Betamethasone; betamethasone acetate phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolotherapy group (Experimental): Subjects randomized to this arm will receive injection(s) of 10% dextrose solution in the affected thumb joint.
  Interventions: Drug: Prolotherapy (10% dextrose solution)
- Corticosteroid Group (Active Comparator): Subjects randomized to this arm will receive injection(s) of betamethasone solution in the affected thumb joint.
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Prolotherapy (10% dextrose solution) — Dextrose diluted with sterile water.
  Arms: Prolotherapy group
Drug: Betamethasone — CELESTONE® SOLUSPAN® * (betamethasone injectable suspension) Injectable Suspension is a sterile aqueous suspension containing 3 mg per milliliter betamethasone, as betamethasone sodium phosphate, and 3 mg per milliliter betamethasone acetate. Subjects will receive a 0.25 to 0.5 mL Celestone Soluspan injection.
  Other Names: Celestone Soluspan
  Arms: Corticosteroid Group

SUMMARY:
Arthritis of the base of the thumb is a common debilitating problem. It is believed that laxity (loosening) of the joint leads to worsening arthritis in this joint. This can be treated by securing the joint surgically or symptoms can be treated with hand therapy and/or injection of corticosteroids. Recently prolotherapy (sugar water) has been shown to decrease looseness of joints and also be helpful for hand and knee arthritis. We hypothesize that prolotherapy injections for thumb arthritis will be equally or more beneficial to the patients than steroids.

DETAILED DESCRIPTION:
Dextrose prolotherapy has been shown to decrease anterior cruciate ligament (ACL) laxity and decrease knee joint pain. Similar to ACL laxity leading to knee osteoarthritis, laxity of the "beak" ligament can lead to worsening thumb CMC osteoarthritis. We hypothesize that dextrose intra-articular prolotherapy will have similar results in treating the pain and instability related to symptomatic thumb CMC osteoarthritis. This will be a prospective randomized double blind comparison study comparing Celestone to Dextrose intra-articular injections as adjuncts to hand therapy for the treatment of symptomatic thumb CMC osteoarthritis. Twenty patients will be randomized to each treatment arm to provide enough power to show a 20% change in visual analogue scale (VAS) for pain to be significant. We will utilize the ultrasound guided injection protocol described by the co-investigators for both treatment arms to ensure proper placement of the respective solutions. We will measure various grip strengths, and VAS pain scales prior to the first injection, prior to the second injection at 6 weeks and at the final visit at 6 months. A telephone follow-up with pain scale will be administered at 3 months. A Quick Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire measuring upper extremity functional impairment will be obtained at initial and final visits.

ELIGIBILITY:
Inclusion Criteria:

* Age >45
* Ability to make follow-up visits over the 6 month protocol
* Ability to give informed consent
* Eaton grade 2-3 thumb carpo-metacarpal joint osteoarthritis with pain over 3/10 on visual analogue scale with symptoms present greater then 6 months.

Exclusion Criteria:

* Recent trauma to the hand or wrist or fractures eeen on radiographs
* Eaton grade 1, or 4 joints affected
* Metabolic bone disease
* Recent systemic or localized infection (within last 2 weeks)
* History of rheumatologic disease
* Allergies to injected solutions
* Thumb carpo-metacarpal joint injections in the prior 6 months.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Gruba, M.D., Principal Investigator — Mayo Clinic Physical Medicine & Rehabilitation Residency
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Asakawa H, Miyagawa J, Higashiyama S, Goishi K, Hanafusa T, Kuwajima M, Taniguchi N, Matsuzawa Y. High glucose and hyperosmolarity increase heparin-binding epidermal growth factor-like growth factor (HB-EGF) production in cultured human aortic endothelial cells. Cell Biochem Funct. 1996 Sep;14(3):181-6. doi: 10.1002/cbf.666. PMID 8888571
- [Background] Berggren M, Joost-Davidsson A, Lindstrand J, Nylander G, Povlsen B. Reduction in the need for operation after conservative treatment of osteoarthritis of the first carpometacarpal joint: a seven year prospective study. Scand J Plast Reconstr Surg Hand Surg. 2001 Dec;35(4):415-7. doi: 10.1080/028443101317149381. PMID 11878178
- [Background] Clarkson MR, Murphy M, Gupta S, Lambe T, Mackenzie HS, Godson C, Martin F, Brady HR. High glucose-altered gene expression in mesangial cells. Actin-regulatory protein gene expression is triggered by oxidative stress and cytoskeletal disassembly. J Biol Chem. 2002 Mar 22;277(12):9707-12. doi: 10.1074/jbc.M109172200. Epub 2002 Jan 9. PMID 11784718
- [Background] Dagenais S, Ogunseitan O, Haldeman S, Wooley JR, Newcomb RL. Side effects and adverse events related to intraligamentous injection of sclerosing solutions (prolotherapy) for back and neck pain: A survey of practitioners. Arch Phys Med Rehabil. 2006 Jul;87(7):909-13. doi: 10.1016/j.apmr.2006.03.017. PMID 16813776
- [Background] Day CS, Gelberman R, Patel AA, Vogt MT, Ditsios K, Boyer MI. Basal joint osteoarthritis of the thumb: a prospective trial of steroid injection and splinting. J Hand Surg Am. 2004 Mar;29(2):247-51. doi: 10.1016/j.jhsa.2003.12.002. PMID 15043897
- [Background] Di Paolo S, Gesualdo L, Ranieri E, Grandaliano G, Schena FP. High glucose concentration induces the overexpression of transforming growth factor-beta through the activation of a platelet-derived growth factor loop in human mesangial cells. Am J Pathol. 1996 Dec;149(6):2095-106. PMID 8952542
- [Background] Glickel SZ. Clinical assessment of the thumb trapeziometacarpal joint. Hand Clin. 2001 May;17(2):185-95. PMID 11478041
- [Background] Hackett, G. (1956). Ligament and Tendon Relaxation Treated by Prolotherapy. Springfield, IL, Charles C Thomas.
- [Background] Han DC, Isono M, Hoffman BB, Ziyadeh FN. High glucose stimulates proliferation and collagen type I synthesis in renal cortical fibroblasts: mediation by autocrine activation of TGF-beta. J Am Soc Nephrol. 1999 Sep;10(9):1891-9. doi: 10.1681/ASN.V1091891. PMID 10477140
- [Background] Jones SC, Saunders HJ, Qi W, Pollock CA. Intermittent high glucose enhances cell growth and collagen synthesis in cultured human tubulointerstitial cells. Diabetologia. 1999 Sep;42(9):1113-9. doi: 10.1007/s001250051279. PMID 10447524
- [Background] Joshi R. Intraarticular corticosteroid injection for first carpometacarpal osteoarthritis. J Rheumatol. 2005 Jul;32(7):1305-6. PMID 15996069
- [Background] Liu YK, Tipton CM, Matthes RD, Bedford TG, Maynard JA, Walmer HC. An in situ study of the influence of a sclerosing solution in rabbit medial collateral ligaments and its junction strength. Connect Tissue Res. 1983;11(2-3):95-102. doi: 10.3109/03008208309004846. PMID 6224646
- [Background] Meenagh GK, Patton J, Kynes C, Wright GD. A randomised controlled trial of intra-articular corticosteroid injection of the carpometacarpal joint of the thumb in osteoarthritis. Ann Rheum Dis. 2004 Oct;63(10):1260-3. doi: 10.1136/ard.2003.015438. PMID 15361383
- [Background] Murphy M, Godson C, Cannon S, Kato S, Mackenzie HS, Martin F, Brady HR. Suppression subtractive hybridization identifies high glucose levels as a stimulus for expression of connective tissue growth factor and other genes in human mesangial cells. J Biol Chem. 1999 Feb 26;274(9):5830-4. doi: 10.1074/jbc.274.9.5830. PMID 10026205
- [Background] Otsuka Y, Mizuta H, Takagi K, Iyama K, Yoshitake Y, Nishikawa K, Suzuki F, Hiraki Y. Requirement of fibroblast growth factor signaling for regeneration of epiphyseal morphology in rabbit full-thickness defects of articular cartilage. Dev Growth Differ. 1997 Apr;39(2):143-56. doi: 10.1046/j.1440-169x.1997.t01-1-00003.x. PMID 9108328
- [Background] Pai S, Talwalkar S, Hayton M. Presentation and management of arthritis affecting the trapezio-metacarpal joint. Acta Orthop Belg. 2006 Jan;72(1):3-10. PMID 16570886
- [Background] Pellegrini VD Jr. Pathomechanics of the thumb trapeziometacarpal joint. Hand Clin. 2001 May;17(2):175-84, vii-viii. PMID 11478040
- [Background] Pugliese G, Pricci F, Locuratolo N, Romeo G, Romano G, Giannini S, Cresci B, Galli G, Rotella CM, Di Mario U. Increased activity of the insulin-like growth factor system in mesangial cells cultured in high glucose conditions. Relation to glucose-enhanced extracellular matrix production. Diabetologia. 1996 Jul;39(7):775-84. doi: 10.1007/s001250050510. PMID 8817101
- [Background] Reeves, K. (2000). Prolotherapy: Basic Science, Clinical Studies, and Technique. Pain Procedures in Clinical Practice. T. A. Lennard. Philadelphia, PA, Hanley and Belfus, INC.: 172-90.
- [Background] Reeves KD, Hassanein K. Randomized prospective double-blind placebo-controlled study of dextrose prolotherapy for knee osteoarthritis with or without ACL laxity. Altern Ther Health Med. 2000 Mar;6(2):68-74, 77-80. PMID 10710805
- [Background] Reeves KD, Hassanein K. Randomized, prospective, placebo-controlled double-blind study of dextrose prolotherapy for osteoarthritic thumb and finger (DIP, PIP, and trapeziometacarpal) joints: evidence of clinical efficacy. J Altern Complement Med. 2000 Aug;6(4):311-20. doi: 10.1089/10755530050120673. PMID 10976977
- [Background] Reeves KD, Hassanein KM. Long-term effects of dextrose prolotherapy for anterior cruciate ligament laxity. Altern Ther Health Med. 2003 May-Jun;9(3):58-62. PMID 12776476
- [Background] Roos MD, Han IO, Paterson AJ, Kudlow JE. Role of glucosamine synthesis in the stimulation of TGF-alpha gene transcription by glucose and EGF. Am J Physiol. 1996 Mar;270(3 Pt 1):C803-11. doi: 10.1152/ajpcell.1996.270.3.C803. PMID 8638660
- [Background] Swigart CR, Eaton RG, Glickel SZ, Johnson C. Splinting in the treatment of arthritis of the first carpometacarpal joint. J Hand Surg Am. 1999 Jan;24(1):86-91. doi: 10.1053/jhsu.1999.jhsu24a0086. PMID 10048521
- [Background] van Beuningen HM, Glansbeek HL, van der Kraan PM, van den Berg WB. Differential effects of local application of BMP-2 or TGF-beta 1 on both articular cartilage composition and osteophyte formation. Osteoarthritis Cartilage. 1998 Sep;6(5):306-17. doi: 10.1053/joca.1998.0129. PMID 10197165
- [Background] Wakitani S, Imoto K, Kimura T, Ochi T, Matsumoto K, Nakamura T. Hepatocyte growth factor facilitates cartilage repair. Full thickness articular cartilage defect studied in rabbit knees. Acta Orthop Scand. 1997 Oct;68(5):474-80. doi: 10.3109/17453679708996266. PMID 9385250
- [Background] Woo SL, Hildebrand K, Watanabe N, Fenwick JA, Papageorgiou CD, Wang JH. Tissue engineering of ligament and tendon healing. Clin Orthop Relat Res. 1999 Oct;(367 Suppl):S312-23. doi: 10.1097/00003086-199910001-00030. PMID 10546655
- [Background] Zhang Y, Niu J, Kelly-Hayes M, Chaisson CE, Aliabadi P, Felson DT. Prevalence of symptomatic hand osteoarthritis and its impact on functional status among the elderly: The Framingham Study. Am J Epidemiol. 2002 Dec 1;156(11):1021-7. doi: 10.1093/aje/kwf141. PMID 12446258

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the pool of referrals to the Mayo Hand Clinic who are interested in receiving an injection for their pain, agree to comply with the standardized hand therapy program, meet the inclusion/exclusion criteria and are able to make the scheduled follow-up visits from Mayo 2008 to July 2010.
Period: Overall Study
Arm/Group | Prolotherapy Group | Corticosteroid Group
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolotherapy Group | Corticosteroid Group | Total
Number analyzed (Participants) | 0 | 2 | 2
Age Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 2 | 2
Gender [Number; unit: participants]
  Female |  | 2 | 2
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decreased Pain Score >20%
Description: Pain was measured on a 10 point visual analogue scale (VAS), with 0 meaning no pain, and 10 meaning extreme pain.
Time Frame: baseline, 6 month follow-up
Arm/Group | Prolotherapy Group | Corticosteroid Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects will be followed for adverse events for six months following the intervention.
Arm/Group | Prolotherapy Group | Corticosteroid Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

LIMITATIONS AND CAVEATS:
Early termination due to low enrollment; no subject data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No